CLINICAL TRIAL: NCT06667232
Title: Evaluating Modulation Effects of Burst Stimulation Patterns Using SEEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-173-002
Record Dates: First submitted 2024-10-27; First posted 2024-10-31 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy
Keywords: burst stimulation patterns; epilepsy; SEEG
MeSH Terms: conditions — Epilepsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single-pulse stimulation (Experimental): Single pulse electrical stimulation (SPES) is an investigational direct electrical stimulation (DES) pattern. Direct cortical stimulation applied at a frequency of ∼1Hz can probe cortico-cortical connections by averaging electrocorticogram time-lock to the stimuli.
  Interventions: Other: Single-pulse stimulation
- Paired-pulse stimulation (Experimental): Paired-pulse stimulation paradigm associates a conditioning and a test stimulation to induce intracortical inhibition or facilitation by modifying the response amplitude.
  Interventions: Other: Paired-pulse stimulation
- Stepwise frequency stimulation (Experimental): Stepwise frequency stimulation is a DES protocol that incrementally increases the stimulation frequency, starting from a lower to higher.
  Interventions: Other: Stepwise frequency stimulation
- Burst stimulation (Experimental): Burst stimulation is a DES patterned repetitive stimulation method; it represents a "more precise" and "smarter" electrical stimulation paradigm. Within a group, high-frequency pulses are emitted, and between groups, low-frequency pulses are delivered. This pattern of pulse delivery more closely mimics the physiological activity of neurons within the brain.
  Interventions: Other: Burst stimulation

INTERVENTIONS:
Other: Single-pulse stimulation — Investigators use single-pulse electrical stimulations at 1Hz to elicit cortico-cortical evoked potentials
  Arms: Single-pulse stimulation
Other: Paired-pulse stimulation — The repetitive delivery of pairs of stimulation pulses is DES patten with a 5-50 ms interval between each pulse, constitutes repetitive paired-pulse stimulation.
  Arms: Paired-pulse stimulation
Other: Stepwise frequency stimulation — Stepwise incremental stimulation ranging from 5 Hz to 145 Hz following a cyclic pattern.
  Arms: Stepwise frequency stimulation
Other: Burst stimulation — Burst stimulation pattern consisting of short bursts delivered once a second and an intraburst frequency of 50 Hz, 100 Hz, 150 Hz, 175 Hz and 200 Hz
  Arms: Burst stimulation

SUMMARY:
The study aims to evaluate modulation effects of burst stimulation patterns via SEEG.

DETAILED DESCRIPTION:
Our research group plans to conduct a study on patients with drug-resistant epilepsy who have SEEG electrodes implanted. The study will evaluate and compare the modulation effect of single-pulse electrical stimulation, paired electrical stimulation, stepwise electrical stimulation, and burst electrical stimulation via direct electrical stimulation using SEEG. The goal is to explore the focal and network modulation effect of distinct stimulation paradigms during the resting state and post-seizure state.

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant focal epilepsy
* Justified SEEG exploration in the context of presurgical assessment of epilepsy
* Subjects will be a part of the epilepsy-monitoring unit for long-term SEEG recordings and analysis
* Written non-opposition to study participation

Exclusion Criteria:

* Pregnant women (Contraindication to SEEG exploration)
* Psychiatric disorders
* History of psychotic disorders
* History of cranial trauma serious (according to the classification), previous or evolutionary other neurological pathology
* Subjects that experience surgical complications during the implant procedure will be excluded from the study

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Modulation Factor | During the trial(up to 3 hours for each subject)
  Investigators calculate normalized the Modulation Factors of single-pulse electrical stimulation, paired electrical stimulation, stepwise electrical stimulation, and burst electrical stimulation patterns using (stimulation-pre-stimulation)/(stimulation + pre-stimulation)
EEG power in spectral frequency bands | During the trial(up to 3 hours for each subject)
  Using SEEG-implanted electrodes, the investigators applied electrical stimulation single-pulse electrical stimulation, paired electrical stimulation, stepwise electrical stimulation, and burst electrical stimulation while observing and recording EEG power changes across six spectral frequency bands during the pre-stimulation, stimulation, and post-stimulation periods.
  EEG Frequency Bands delta (1-4 Hz) theta (5-8 Hz) alpha (9-12 Hz) beta (13-30 Hz) low gamma (31-70 Hz) high gamma (71-150 Hz)
Phase Locking Value | During the trial(up to 3 hours for each subject)
  To estimate functional connectivity through the oscillatory synchrony of two brain regions, phase locking value (PLV) provides a measure of inter-regional synchrony based on phase difference between the paired signals.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China